CLINICAL TRIAL: NCT01484067
Title: A Randomized, Clinician-Blind, Clinical Study to Examine the Safety and Performance of Compeed© Total Care™ Cold Sore Patch With Zinc Sulfate for the Treatment of Herpes Labialis
Brief Title: Study of a Cold Sore Patch for the Treatment of Herpes Labialis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Products Company Division of Johnson & Johnson Consumer Companies, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCOWDH0003; 44-DRM-HLS-11-002 (Other: CRO)
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Herpes Labialis
Keywords: Herpes Simplex Virus
MeSH Terms: conditions — Herpes Labialis; Herpes Simplex | interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patch (Experimental): At onset of signs/symptoms, subjects will apply assigned patch, and return to study center within 24 hours. Patch will be worn continuously, being replaced as needed.
  Interventions: Device: Patch ( Compeed© Total CareTM Cold Sore Patch)
- No Patch (No Intervention): No treatment will be initiated at onset of signs and symptoms although subject is still required to return to study center with 24 hours of onset of signs/symptoms.

INTERVENTIONS:
Device: Patch ( Compeed© Total CareTM Cold Sore Patch) — A cold sore patch containing zinc sulfate
  Other Names: Compeed© Total CareTM Cold Sore Patch
  Arms: Patch

SUMMARY:
If a person qualifies to participate in this study, they will have an equal chance of being assigned to either of two groups. One group will receive a patch that they will need to carry with them, because as soon as a cold sore starts (within 1 hour) they will need to put the patch over the sore. The other group will not get a patch, but will need to follow the other instructions anyway.

When a subject's outbreak begins, they will need to return to the study center within 24 hours. Then they will return according to the appointments given within 10 days. If the study staff sees that their sore has healed enough before 10 days, subjects will be told that they don't need to return again.

As long as subjects are in the study, they will need to answer a few simple questions every day on a card or booklet called a diary, starting the first day of their outbreak. If a subject is assigned to the patch group, they must wear the patch all the time, taking it off only to replace it (if it gets loose, dirty, or unsightly) and at the study center, when they are asked to remove the patch so the sore can be checked.

During the study subjects will be allowed to use paracetamol for pain, but no other treatments or medicine. If they use paracetamol, subjects must record it in their diary. The study will be stopped, and there will be no subject visits or treatments during the end of year holiday break. If a subject experiences an outbreak during the holiday, they may follow their usual treatment routine.

DETAILED DESCRIPTION:
This is a two-arm, randomized, clinician-blind study. No severe adverse effects are expected to be experienced in the control group. All subjects are allowed to treat cold sore related pain with an oral analgesic - paracetamol (APAP). The use of APAP for pain will be recorded as a concomitant medication. However, subjects will be required to refrain from using any additional treatment (topical or systemic) during study participation.

Subjects randomized to treatment will be instructed to initiate the therapy within 1 hour onset of their first sign or symptom and record their assessment in the diary card (for no treatment subjects, they will only record assessments upon onset of first sign or symptom). All subjects will return to the study center for clinical assessments within 24 hours and 48 hours after onset of first sign or symptom/initiation of treatment and every other day thereafter, with a final visit at Day 10 or at the time of completion/discontinuation if before Day 10. Diaries will be completed each day, beginning upon initiation of therapy (Day 0) and continuing until study completion/discontinuation, and will include information on study product applications.

Subjects assigned to a patch treatment will wear a patch continuously on their lesion and will apply a new patch on occasions where the patch becomes loose, falls off or becomes unsightly, including at study visits to the facility where subjects will be asked to remove their patch for clinical assessments. Treatment will continue until the lesion is healed, for a maximum of 10 days. As the test period will possibly extend through the end of year holiday break, subject visits and treatments will be halted during this break. All subjects who have not initiated therapy including subjects assigned no treatment group, will be allowed to use their regular therapy for a cold sore outbreak during the holiday break.

ELIGIBILITY:
Inclusion Criteria:

* Female or male 18-70 years old in good general health
* Has a history of Herpes Labialis in the areas and with the frequency defined in the protocol.
* Based on history, likely to experience a cold sore outbreak within next 2 to 3 months
* Willing to provide informed consent
* Willing to stop all other treatment of this condition and any topical products (lip balm, cosmetics, sunscreen) during test period
* Women of child bearing potential must agree to use an adequate method of birth control (systemic birth control/intrauterine device)

Exclusion Criteria:

* Self-reported to be pregnant, planning to become pregnant or nursing
* Has any medical history or condition that might, per protocol or in the opinion of the investigator, compromise the subject's safety or the analysis of results.
* Is taking or has taken within the 28 days before commencing treatment, protocol-specified medications or herbal supplements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Overall Condition of Cold Sore | Within 10 Days
  Taking into account the size, physical impression of the lesion and overall quality of healing, clinician will score the overall condition of the cold sore on a scale of 0-10, where 0=Best and 10=Worst.
Erythema | Within 10 Days
  Clinician's score on a scale of 0-10 for erythema, where 0=none and 10=most severe
Edema | Within 10 Days
  Clinician's score on a scale of 0-10 for edema, where 0=none and 10=most severe
Vesicles | Within 10 Days
  Clinician's score on a scale of 0-10 for vesicles, where 0=none and 10=most severe
Scab/Crust | Within 10 Days
  Clinician's score on a scale of 0-10 for scab/crust, where 0=none and 10=most severe

SECONDARY OUTCOMES:
Lesion Size | Within 10 Days
  Measurement of lesion diameter
Lesion Stage | Within 10 Days
  Lesion Stage on a categorical scale of 1-8, as described below:
  1. = prodrome (symptoms including itching, pain, tingling, but no physical evidence of disease by inspection or by palpation)
  2. = maculae (erythema)
  3. = papule (any elevation of skin without fluid; solid raised lesion)
  4. = vesicle (blister, fluid filled or collapsed)
  5. = ulcer/eroson (moist sore/wound)
  6. = soft crust/scab
  7. = hard crust/scab
  8. = healed (normal skin with no signs or symptoms; residual postlesion skin changes such as erythema, flaking, or slight asymmetry may be present)
Pain | Within 10 Days
  Subject's score for unprovoked pain on a scale of 0-10, where 0=none and 10=most severe
Discomfort | Within 10 Days
  Subject's score for discomfort on a scale of 0-10, where 0=none and 10=most severe
Itching | Within 10 days
  Subject's score for itching on a scale of 0-10, where 0=none and 10=most severe
Burning | Within 10 Days
  Subject's score for burning on a scale of 0-10, where 0=none and 10=most severe
Tingling | Within 10 Days
  Subject's score for tingling on a scale of 0-10, where 0=none and 10=most severe
Swelling | Within 10 Days
  Subject's score for swelling on a scale of 0-10, where 0=none and 10=most severe
Soreness/Tenderness | Within 10 Days
  Subject's score for soreness/tenderness [upon touching] on a scale of 0-10, where 0=none and 10=most severe
Redness | Within 10 Days
  Subject's score for redness on a scale of 0-10, where 0=none and 10=most severe
Blisters | Within 10 Days
  Subject's score for blisters on a scale of 0-10, where 0=none and 10=most severe
Scab or Crust | Within 10 Days
  Subject's score for scab or crust on a scale of 0-10, where 0=none and 10=most severe

CONTACTS AND LOCATIONS:
Overall Officials: Clare Kendall, Study Director — Johnson & Johsnon Consumer and Personal Products Worldwide
Locations (1):
- Intertek CRS, Manchester, United Kingdom